CLINICAL TRIAL: NCT00328952
Title: Naturalistic Multicenter Study of Changes in Auditory Verbal Hallucination During Atypical Antipsychotic Treatment of Schizophrenia
Brief Title: Changes in Auditory Verbal Hallucination During Atypical Antipsychotic Treatment of Patients With Schizophrenia
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Collaborators: Hallym University Medical Center (Other); Gachon University Gil Medical Center (Other)
Responsible Party: Yong Min Ahn/Associate Professor, Seoul National University Hospital
Other Study IDs: KYS-2006-05018
Record Dates: First submitted 2006-05-22; First posted 2006-05-24 (Estimated); Last update posted 2009-09-16 (Estimated); Status verified 2009-09

CONDITIONS: Schizophrenia; Hallucinations
Keywords: schizophrenia; auditory verbal hallucination; antipsychotic treatment
MeSH Terms: conditions — Schizophrenia; Hallucinations

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — routine lab tests for changes in medical condition
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to evaluate the changes in various aspects of auditory verbal hallucinations during 24-week antipsychotic treatment in naturalistic condition.

DETAILED DESCRIPTION:
Auditory verbal hallucinations (AVH), meaning the experience of hearing voices, occur in 60-75% of patients with schizophrenia. Patients experiencing persistent AVH tend to be interrupted in their daily routines and have trouble keeping regular jobs due to the intrusiveness or abusive contents of voices. In addition, auditory hallucinations are reported to remain even after disappearance of other psychotic symptoms in many patients with schizophrenia spectrum disorders after treatment with typical antipsychotics.

The study involves detailed phenomenological assessments of AVH and other psychotic symptoms, as well as side effects of atypical antipsychotics.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients, 15-65 years of age
* Patients must have a diagnosis of schizophrenia according to the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV)>
* Patients experiencing vivid AVH confirmed by score of 4 or above using hallucinatory behavior item on Positive And Negative Syndrome Scale (PANSS).
* Patients who are drug-naive or drug-free for more than 4 weeks.
* Patients who are scheduled to receive atypical antipsychotic medication.
* Each patient must provide written informed consent after full explanation of study protocol, and authorized legal guardian must understand the nature of the study and must also give assent to study participation.
* Subjects who are fluent in Korean.

Exclusion Criteria:

* DSM-IV substance (except nicotine or caffeine) dependence within the past 1 year.
* Mental retardation (IQ < 70).
* Neurological disorders including epilepsy, stroke, or severe head trauma.
* Clinically significant laboratory abnormalities, on any of the following tests: CBC with differential, electrolytes, BUN, creatinine, hepatic transaminases, urinalysis and EKG.
* Treatment with an injectable depot neuroleptic within less than three dosing interval between the last depot neuroleptic injections and baseline.
* History of electroconvulsive therapy or transcranial magnetic stimulation within the past 3 months.
* Subjects who are not fluent in Korean.

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: voice-hearing patients with schizophrenia
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2004-08; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jong-Hoon Kim, MD, PhD, Study Director — Gachon University Gil Medical Center; Jung Seo Yi, MD, PhD, Study Director — Hallym University Medical Center
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Background] Shergill SS, Murray RM, McGuire PK. Auditory hallucinations: a review of psychological treatments. Schizophr Res. 1998 Aug 17;32(3):137-50. doi: 10.1016/s0920-9964(98)00052-8. PMID 9720119
- [Background] Farhall J, Gehrke M. Coping with hallucinations: exploring stress and coping framework. Br J Clin Psychol. 1997 May;36(2):259-61. doi: 10.1111/j.2044-8260.1997.tb01411.x. PMID 9167865
- [Background] Haddock G, McCarron J, Tarrier N, Faragher EB. Scales to measure dimensions of hallucinations and delusions: the psychotic symptom rating scales (PSYRATS). Psychol Med. 1999 Jul;29(4):879-89. doi: 10.1017/s0033291799008661. PMID 10473315
- [Background] Nayani TH, David AS. The auditory hallucination: a phenomenological survey. Psychol Med. 1996 Jan;26(1):177-89. doi: 10.1017/s003329170003381x. PMID 8643757
- See also: Click here for the information about approaches to hallucination control in schizophrenia. — http://www.schizophrenia.com/schizoph/hallucontrol.html